CLINICAL TRIAL: NCT05236634
Title: Comparative Study Between Fixed Dose Monotherapy (Phosphodiesterase 5 Inhibitors or Alpha Blockers) Versus Combined Therapy in Benign Prostatic Hyperplasia Patients With Lower Urinary Tract Symptoms
Brief Title: (Phosphodiesterase 5 Inhibitors & α-blockers): Single Versus Combined Therapy in Benign Prostatic Hyperplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Hussein Mostafa, Principle Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Drug therapies in BPH
Record Dates: First submitted 2022-01-14; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Phosphodiesterase5 inhibitors and Alpha Blockers
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Phosphodiesterase 5 Inhibitors; Tadalafil; Tablets; Adrenergic alpha-Antagonists

STUDY DESIGN:
Intervention Model Description: A total of (120) patients with LUTS due to BPH fulfilling the inclusion criteria will be included in this study. Patients will be randomly divided into 3 groups: Group A: Forty patients with LUTS due to BPH will be given tamsulosin 0.4 mg for 12 weeks. Group B: Forty patients with LUTS due to BPH will be given tadalafil 5 mg for 12 weeks. Group C: Forty patients with LUTS due to BPH will be given combined therapy for 12 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Active Comparator): Forty patients with LUTS due to BPH will be given tamsulosin 0.4 mg for 12 weeks.
  Interventions: Drug: Alpha Blockers
- Group B (Active Comparator): Forty patients with LUTS due to BPH will be given tadalafil 5 mg for 12 weeks.
  Interventions: Drug: Phosphodiesterase 5 Inhibitors
- Group C (Active Comparator): Forty patients with LUTS due to BPH will be given combined therapy(tamsulosin 0.4 mg and tadalafil 5 mg) for 12 weeks.
  Interventions: Drug: Combined Alpha Blockers and Phosphodiesterase 5 Inhibitors

INTERVENTIONS:
Drug: Phosphodiesterase 5 Inhibitors — A total of (120) patients with LUTS due to BPH fulfilling the inclusion criteria will be included in this study. Patients will be randomly divided into three groups: Group A: Forty patients with LUTS due to BPH will be given tamsulosin 0.4 mg for 12 weeks. Group B: Forty patients with LUTS due to BPH will be given tadalafil 5 mg for 12 weeks. Group C: Forty patients with LUTS due to BPH will be given combined therapy for 12 weeks.
  Other Names: tadalafil 5 mg oral Tablet
  Arms: Group B
Drug: Alpha Blockers — A total of (120) patients with LUTS due to BPH fulfilling the inclusion criteria will be included in this study. Patients will be randomly divided into three groups: Group A: Forty patients with LUTS due to BPH will be given tamsulosin 0.4 mg for 12 weeks. Group B: Forty patients with LUTS due to BPH will be given tadalafil 5 mg for 12 weeks. Group C: Forty patients with LUTS due to BPH will be given combined therapy for 12 weeks.
  Other Names: Tamsulin 0.4 mg oral tablet
  Arms: Group A
Drug: Combined Alpha Blockers and Phosphodiesterase 5 Inhibitors — A total of (120) patients with LUTS due to BPH fulfilling the inclusion criteria will be included in this study. Patients will be randomly divided into three groups: Group A: Forty patients with LUTS due to BPH will be given tamsulosin 0.4 mg for 12 weeks. Group B: Forty patients with LUTS due to BPH will be given tadalafil 5 mg for 12 weeks. Group C: Forty patients with LUTS due to BPH will be given combined therapy for 12 weeks.
  Other Names: Tadalafil 5 mg oral Tablet and Tamsulin 0.4 mg oral tablet
  Arms: Group C

SUMMARY:
To compare between efficacy of phosphodiesterase5 inhibitors (tadalafil 5 mg) and Alpha Blockers (tamsulosin 0.4 mg) monotherapy vs combined therapy in treatment of lower urinary tract symptoms of benign prostatic hyperplasia.

DETAILED DESCRIPTION:
The proposed research aims to answer the question about efficacy and safety of phosphodiesterase 5 inhibitors (tadalafil 5 mg) and Alpha Blockers (tamsulosin 0.4 mg) monotherapy vs combined therapy in treatment of lower urinary tract symptoms of benign prostatic hyperplasia .

Benign prostatic hyperplasia (BPH) is a disorder histologically characterized as the non-malignant hyperplasia of prostatic cells. Most of patients with BPH present with lower urinary tract symptoms (LUTS). About half of men develop BPH, among those; about half develop some degree of bladder outlet obstruction (BOO). BOO and/or changes in smooth muscle tone and resistance that can accompany BPH may result in (LUTS).

Alpha-blockers have been widely used for the treatment of LUTS/BPH for a long time. Some alpha-blockers may cause ejaculatory dysfunction in some individuals. Tadalafil, a (PDE-5), was approved by the Food and Drug Administration (FDA) for the treatment of (ED) in 2003 and for the treatment of BPH in 2011.

The PDE5 inhibitors are used in the treatment of ED and there are increasing data of effects of these drugs on bladder and urethral relaxation as well as of prostatic smooth muscles that may relief the symptoms of BPH.

Medical treatments for LUTS/BPH are able to significantly impact on sexual function. Sexual side effects like ejaculatory dysfunction, reduced or lost libido, and ED have been widely reported in patients treated with alpha blockers (ABs) and 5-alpha reductase inhibitors, the most utilized drugs for the treatment of LUTS/BPH.

The inclusion of Tadalafil in complex of combined conservative therapy of patients with BPH not only improves sexual function but has a positive effect on symptoms of the disease and the psychological state of the patient.

ELIGIBILITY:
Inclusion Criteria:

1 - Men > 45 years with LUTS/BPH for > 6 months 2- IPSS of ≥ 8 and Qmax of ≥ 4 to≤ 15 mL/s

Exclusion Criteria:

1. PSA level of > 10.0 ng/mL (if ≥ 4.0 to≤ 10.0 ng/mL prostate cancer will be excluded).
2. Post-voidresidual urine volume of ≥ 150 mL.
3. Previous Urine Retention or Urethral Catheterization .
4. other pathology such as urinary bladder stone , bladder mass or neurogenic bladder .
5. Any case of LUTS other than BPH (urinary bladder stone, neurogenic bladder, bladder neck contracture,rethral stricture, bladder cancer, acute or chronic prostatitis, acute or chronic urinary tract infection).
6. patients supposed to undergo intraocular operation (as cataract operation) .
7. History of head injury or cerebrovascular stroke or spinal injury.
8. pelvic fracture.
9. Uncontrolled diabetic patient.
10. Patients with chronic obstructive lung disease on medical treatment.
11. Parasympatholytic drugs are contraindicated during the study. 12. Patients refusing to share in the study.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men > 45 years
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in International prostate symptom score (IPSS) after 12 weeks | At start of study and after 12 weeks from drug intake
  The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Change in International index of erectile function (IIEF) after 12 weeks | At start of study and after 12 weeks from drug intake
  The International Index of Erectile Function (IIEF) is a widely used, multi-dimensional self-report instrument for the evaluation of male sexual function. It is has been recommended as a primary endpoint for clinical trials of erectile dysfunction (ED) and for diagnostic evaluation of ED severity.
Change in Maximal urinary flow rate (Qmax) after 12 weeks | At start of study and after 12 weeks from drug intake
  The flow rate is calculated as milliliters (ml) of urine passed per second. Both average and top flow rates are measured. The fastest flow rate, also known as Qmax, is used to understand if a block or obstruction is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Osman, MD, Study Chair — Assiut University, Urology department, Faculty of Medicine

REFERENCES:
- [Background] Singh DV, Mete UK, Mandal AK, Singh SK. A comparative randomized prospective study to evaluate efficacy and safety of combination of tamsulosin and tadalafil vs. tamsulosin or tadalafil alone in patients with lower urinary tract symptoms due to benign prostatic hyperplasia. J Sex Med. 2014 Jan;11(1):187-96. doi: 10.1111/jsm.12357. Epub 2013 Oct 25. PMID 24165272
- [Background] Wang XH, Wang X, Shi MJ, Li S, Liu T, Zhang XH. Systematic review and meta-analysis on phosphodiesterase 5 inhibitors and alpha-adrenoceptor antagonists used alone or combined for treatment of LUTS due to BPH. Asian J Androl. 2015 Nov-Dec;17(6):1022-32. doi: 10.4103/1008-682X.154990. PMID 25994648
- [Background] Mirone V, Sessa A, Giuliano F, Berges R, Kirby M, Moncada I. Current benign prostatic hyperplasia treatment: impact on sexual function and management of related sexual adverse events. Int J Clin Pract. 2011 Sep;65(9):1005-13. doi: 10.1111/j.1742-1241.2011.02731.x. Epub 2011 Jul 1. PMID 21718399
- See also: Gravas S, Cornu JN, Gacci M, Gratzke C, Herrmann TR, Mamoulakis C, Rieken M, Speakman MJ and Tikkinen KA. (2015): Guidelines on the management of non neurogenic male (LUTS), incl. (BPO). EAU Guidelines — https://uroweb.org/guideline/treatment-of-non-neurogenic-male-luts/#1
- See also: Gravas S, Cornu JN, Gacci M, Gratzke C, Herrmann TRW, Mamoulakis C, et al. Management of nonneurogenic male LUTS. In: EAU Guidelines 2020. Arnhem,The Netherlands: EAU Guidelines Office; 2020. Available from:https://uroweb.org/guideline/treatment-of-non — https://uroweb.org/guideline/treatment-of-non-neurogenic-male-luts/.